CLINICAL TRIAL: NCT05654831
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Repeated Dose Escalation, First-Time-In-Human Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ECC5004 in Healthy Participants and in Patients With Type 2 Diabetes Mellitus
Brief Title: FTIH of ECC5004 in Healthy and Diabetic Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eccogene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: EC0004
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAD Cohorts 1 to 2: Participants receiving Placebo (Placebo Comparator): Participants in each SAD cohort will be randomized to receive placebo.
  Interventions: Drug: Placebo
- SAD Cohorts 1 to 2: Participants receiving ECC5004 (Experimental): Participants in each SAD cohort will be randomized to receive up to 4 escalating doses of ECC5004 ranging from 1 mg to 300 mg.
  Interventions: Drug: ECC5004
- MAD Cohorts 1 to 4: Participants receiving Placebo (Placebo Comparator): Participants will be randomized to receive a once-daily dose of placebo for 28 days.
  Interventions: Drug: Placebo
- MAD Cohorts 1 to 4: Participants receiving ECC5004 (Experimental): Participants will be randomized to receive a once-daily dose of 1 of 4 escalating doses of ECC5004 ranging from 10 mg to 150 mg for 28 days.
  Interventions: Drug: ECC5004

INTERVENTIONS:
Drug: Placebo — Matching Placebo will be administered as oral tablet. Matching Placebo will be given orally during each dosing day.
  Arms: MAD Cohorts 1 to 4: Participants receiving Placebo; SAD Cohorts 1 to 2: Participants receiving Placebo
Drug: ECC5004 — ECC5004 will be administered as oral tablet(s) during each dosing day.
  Arms: MAD Cohorts 1 to 4: Participants receiving ECC5004; SAD Cohorts 1 to 2: Participants receiving ECC5004

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose and multiple ascending dose study of ECC5004 in healthy participants and in patients with Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
This study will be conducted in two cohorts of Single Ascending Dose (SAD) with a dose range from 1mg to 300mg, and in four cohorts of Multiple Ascending Dose (MAD) with a dose range of 10mg to 150mg to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ECC5004 in Healthy Participants and in Patients with Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants of non-childbearing potential
* Age of 18 to 65 years
* BMI of 18.0 to 32.0 kg/m2
* Hemoglobin A1c ≤ 6.0%
* Female participants who are postmenopausal, confirmed by FSH test, or surgically sterile, confirmed by medical documentation, or agree to practice true abstinence
* Male participants agree to use contraception, or agree to practice true abstinence
* No clinically significant findings in physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, laboratory tests, or medical/psychiatric history
* Able to understand and sign and date informed consent

Additional Inclusion Criteria for Part 2 (MAD)

* Diagnosed Type 2 Diabetes Mellitus of 18 to 70 years of age inclusive
* Type 2 Diabetes Mellitus with lifestyle modification only or with stable dose of metformin for ≥ 2 months prior to the study treatment
* BMI of 24.0 to 40.0 kg/m2 with a minimum body weight of 50.0 kg (110 lbs)
* HbA1c ≥ 7.0% and ≤ 10.5%, and fasting plasma glucose ≤ 270 mg/dL
* Blood pressure (BP) with or without medication: Systolic BP ≤ 160 mmHg, AND Diastolic BP ≤ 100 mmHg
* Not taking any active treatment regimen

Exclusion Criteria:

* Concomitant participation in any investigational study of any nature
* Blood loss of non-physiological reasons ≥ 200 ml (i.e. trauma, blood collection, blood donation) within 2 months prior to the first dose of study drug, or plan to donate blood during this trial and within 1 month after the last dosing
* Unable to refrain from taking any non-metformin anti-diabetic medication including insulin within ≥ 3 months prior to the study treatment
* Serum calcitonin > 20 ng/L
* Clinically relevant acute or chronic medical conditions or diseases of the cardiovascular, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, psychiatric, immune or dermatologic systems
* Diagnosis of T1DM or secondary forms of diabetes
* Individual or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia 2 (MEN2), or suspected MTC
* History of pancreatitis
* Significant allergic reaction to active ingredients or excipients of the study drug.
* Any clinically significant abnormal findings in the participant's physical examination, laboratory tests, pregnancy test, urine drug screen, alcohol test, or medical history which in the opinion of the Investigator would prevent the participants from participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events, with abnormal laboratory test results, abnormal ECGs, abnormal vital signs, and abnormal physical examinations | SAD: Up to Day 8 and MAD: Up to Day 35
  Safety Assessment evaluated through adverse events, laboratory evaluations, vital signs, ECGs, and physical examination.

SECONDARY OUTCOMES:
Pharmacokinetic Parameters: AUC0-24 | SAD: Up to Day 3 and MAD: Up to Day 30
  AUC from time 0 to 24 hour dosing interval
Pharmacokinetic Parameters: AUC0-tlast | SAD: Up to Day 3
  AUC from time 0 to the time of last quantifiable non-zero concentration
Pharmacokinetic Parameters: AUC0-tau | MAD: Up to Day 30
  AUC over a dosing interval from time 0 to time of last quantifiable concentration
Pharmacokinetic Parameters: AUC0-infinity | SAD: Up to Day 3
  AUC from time 0 extrapolated to infinity
Pharmacokinetic Parameters: Cmax | SAD: Up to Day 3 and MAD: Up to Day 30
  Maximum observed plasma concentration
Pharmacokinetic Parameters: C24 | SAD: Up to Day 3 and MAD: Up to Day 30
  Observed concentration at 24 hours post dose
Pharmacokinetic Parameters: Ctau | MAD: Up to Day 30
  Observed concentration at the end of the dosing interval
Pharmacokinetic Parameters: tmax | SAD: Up to Day 3 and MAD: Up to Day 30
  Time of the maximum observed plasma concentration
Pharmacokinetic Parameters: tlag | SAD: Up to Day 3 and MAD: Up to Day 30
  Lag time (time delay between dosing and first observed plasma concentration)
Pharmacokinetic Parameters: t1/2 | SAD: Up to Day 3 and MAD: Up to Day 30
  Apparent terminal elimination half-life
Pharmacokinetic Parameters: Clast | SAD: Up to Day 3
  Last measurable non-zero concentration
Pharmacokinetic Parameters: tlast | SAD: Up to Day 3
  Time of last measurable non-zero concentration
Pharmacokinetic Parameters: CL/F | SAD: Up to Day 3 and MAD: Up to Day 30
  Apparent Clearance
Pharmacodynamic Parameters: AUC0-4 for glucose | MAD: Up to Day 30
  AUC from time 0 to 4 hour dosing interval
Pharmacodynamic Parameters: AUC0-4 for insulin | MAD: Up to Day 30
  AUC from time 0 to 4 hour dosing interval
Pharmacodynamic Parameters: AUC0-4 for glucagon | MAD: Up to Day 30
  AUC from time 0 to 4 hour dosing interval
Pharmacodynamic Parameters: AUC0-4 for C-peptide | MAD: Up to Day 30
  AUC from time 0 to 4 hour dosing interval
Pharmacodynamic Parameters: Fasting plasma glucose | MAD: Up to Day 30
  Change from baseline
Pharmacodynamic Parameters: Mean daily glucose | MAD: Up to Day 30
  Change from baseline
Pharmacodynamic Parameters: Body Weight and Waist Circumference | MAD: Up to Day 30
  Change from baseline
Pharmacodynamic Parameters: Fasting plasma glucose homeostatic model assessment | MAD: Up to Day 30
  Fasting plasma glucose homeostatic model assessment
Pharmacodynamic Parameters: Fasting plasma insulin homeostatic model assessment | MAD: Up to Day 30
  Fasting plasma insulin homeostatic model assessment

CONTACTS AND LOCATIONS:
Overall Officials: Eccogene, Study Director — Eccogene Clinical Trials
Locations (1):
- Eccogene Investigational Site, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haggag AZ, Xu J, Butcher L, Pagnussat S, Davies G, Lundqvist S, Wang W, Van Zuydam N, Nelander K, Jha A, Yu H, Boianelli A, Lindmark B, Ollerstam A, Sun X, Wang F, Pan X, Liu H, Chen W, Xu J, Wallenius K, Zhou J. Non-clinical and first-in-human characterization of ECC5004/AZD5004, a novel once-daily, oral small-molecule GLP-1 receptor agonist. Diabetes Obes Metab. 2025 Feb;27(2):551-562. doi: 10.1111/dom.16047. Epub 2024 Nov 4. PMID 39495140